CLINICAL TRIAL: NCT03157115
Title: Validation of Kinocardiography, New Technology for Cardiac Linear and Torsional Contractility Measurement, to Assess Heart Failure Patient With Low Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Dr Marielle Morissens, MD, Brugmann University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHUB-Kino-HFrEF
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Impaired Left Ventricular Ejection Fraction
Keywords: Kinocardiography; Cardiac contractility; Heart kinetic energy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Impaired left ventricular ejection fraction (Experimental): Patients with reduced left ventricular ejection fraction (< 50 %)
  Interventions: Device: Kinocardiography
- Control (Active Comparator): Patients with a normal left ventricular ejection fraction (≥ 50 %), without heart failure. The patients from the reduced left ventricular ejection fraction group will be matched with patients from the control group for sex, age, BMI and cardiovascular treatment.
  Interventions: Device: Kinocardiography

INTERVENTIONS:
Device: Kinocardiography — This device records the electric and mechanic function of the heart. With electrodes and adequate electronics, ECG is recorded. 6 degrees of freedom accelerometers are also included in the device to measure the micro accelerations of the body at the body surface when the device is placed on the skin. Using physics principles and adequate calibration, those accelerations allow us to calculate parameters such as kinetics energies related to cardiac contractility.
  During a standard echocardiography appointment for a patient suffering from a cardiovascular condition with/without heart failure, the cardiologist will monitor the heart of the patient with the Kino device (examination lasting a few minutes with the patient lying down on a bed). Data will be matched between the control group and the experimental group.

SUMMARY:
Measuring cardiac contractility is commonly realized with gold standard echocardiography or MRI. Portable devices to measure this contractility are not available as for rhythm and electric function assessment. The new Kinocardiography technology could provide a non invasive and portable tool to measure contractility.

This device records the electric and mechanic function of the heart simultaneously. With electrodes and adequate electronics, ECG is recorded. 6 degrees of freedom accelerometers are also included in the device to measure the micro accelerations of the body at the body surface when the device is placed on the skin. Using physics principles and adequate calibration, those accelerations allow the investigators to calculate parameters such as kinetics energies related to cardiac contractility. Kinocardiography is a non invasive and portable technology.

ELIGIBILITY:
Inclusion Criteria:

* Control group: Left Ventricle Ejection Fraction ≥ 50 %
* Heart failure patients: Left Ventricle Ejection Fraction < 50 %

Exclusion Criteria:

* Intracardiac devices and arrhythmia at the time of assessment
* Participates in other clinical study or trial.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Total heart kinetic energy | 1 hour
  Computed according to the micro accelerations of the body at the body surface. The hypothesis is that the investigators will observe a lower total heart kinetic energy for the group with impaired left ventricular ejection fraction in comparison to a paired control patient group.

SECONDARY OUTCOMES:
Ratio of torsional kinetic energy over total kinetic energy | 1 hour
  Computed according to the micro accelerations of the body at the body surface. The hypothesis is that the investigators will observe a lower ratio of torsional kinetic energy over total kinetic energy for the impaired left ventricular ejection fraction group in comparison to a paired control group.

CONTACTS AND LOCATIONS:
Overall Officials: Eva De Keyzer, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Keyzer E, Hossein A, Rabineau J, Morissens M, Almorad A, van de Borne P. Non-invasive cardiac kinetic energy distribution: a new marker of heart failure with impaired ejection fraction (KINO-HF). Front Cardiovasc Med. 2023 May 2;10:1096859. doi: 10.3389/fcvm.2023.1096859. eCollection 2023. PMID 37200972